CLINICAL TRIAL: NCT04084717
Title: Phase II Study of Crizotinib for ROS1 and MET Activated Lung Cancer (CROME)
Brief Title: Study of Crizotinib for ROS1 and MET Activated Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-5607; CROME / WI235747 (Other: Princess Margaret Cancer Centre)
Record Dates: First submitted 2019-09-08; First posted 2019-09-10 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Non-squamous Non-small-cell Lung Cancer; Stage IV Non-small Cell Lung Cancer; ROS1 Gene Rearrangement; MET Activating Mutation; MET Amplification
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of the following:
  Cohort 1 - ROS1 rearrangement Cohort 2 - MET-activating mutation (exon 14) Cohort 3 - MET-amplification
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ROS1 Rearrangement (Experimental): Patients with stage IV or incurable non-squamous non-small cell lung cancer with a documented ROS1 rearrangement will be assigned to this arm.
  Interventions: Drug: Crizotinib
- MET-activating Mutation (exon 14) (Experimental): Patients with stage IV or incurable non-squamous non-small cell lung cancer with a documented MET-activating mutation (exon 14) will be assigned to this arm.
  Interventions: Drug: Crizotinib
- MET-amplification (Experimental): Patients with stage IV or incurable non-squamous non-small cell lung cancer with a documented MET-amplification will be assigned to this arm.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — Crizotinib is an orally administered, chemotherapy drug that works by blocking ALK, MET and ROS1 receptor tyrosine kinases from working.
  Participants will receive crizotinib, orally (by mouth), at a dose of 250 mg, twice per day, every day of each 28 day cycle.
  Other Names: XALKORI

SUMMARY:
This is a phase 2 study of a drug called crizotinib in people with metastatic (the cancer has spread to other parts of the body) non-small cell lung cancer with a mutation (change) in genes called ROS1 or MET. The purpose of this study is to look at how effective crizotinib is at treating ROS1 or MET mutated non-small cell lung cancer.

Crizotinib, also called XALKORI, is a chemotherapy drug that is currently approved for the treatment of ALK- or ROS1- positive advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
The study consists of a screening period, study drug period, end of study drug visit and follow-up period.

During the screening period, participants will be asked to have tests and procedures done to make sure that they are eligible to continue in the study. Screening may take several visits. Participants found to be eligible to continue in the study, will then enter the study drug period where they will take the study drug and have tests and procedures done about once a week for safety and for research purposes.

Participants who stop the study drug completely for any reason, will be asked to return to the clinic for an end of study drug visit about 28 days after their last dose of study drug to have tests and procedures done for safety and for research purposes. Participants that are experiencing any side effects during this time, will be closely followed by their study Doctor until the side effects have resolved or stabilized.

Participants who discontinue study drug for any reason other than disease progression, will be asked to have radiological imaging every 8 weeks to follow up on the status of their disease, until disease progression or the start a new treatment for their cancer.

After their final visit, the study nurse will call participants approximately every 3 months to check on the status of their health.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of stage IV or incurable non-squamous non-small cell lung cancer with a documented ROS1 rearrangement (cohort 1) or MET-activating mutation (exon 14) (cohort 2) or MET-amplification (cohort 3) tested in either plasma or tissue, as applicable
* 18 years of age or older.
* Measurable disease as per RECIST v1.1.
* Adequate hematologic and organ function within 7 days of the proposed start date of treatment and adequate cardiac function within 28 days of the proposed start date of treatment
* Life expectancy >12 weeks.
* Have the ability to understand and the willingness to sign a written informed consent document
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* No contraindication to Crizotinib therapy
* Able to swallow and retain oral medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* No pregnant
* Agree to use methods (as agreed upon by the study doctor and participant) before the study and for at least 120 days after the last dose of study drug to prevent pregnancy

Exclusion Criteria:

* Symptomatic untreated brain metastases.
* Had chemotherapy (including investigational cytotoxic chemotherapy), biologic agents (e.g. targeted therapy or antibodies) within 4 weeks or radiotherapy within 2 weeks prior to the proposed first dose of study treatment.
* Adverse events attributed to prior anti-cancer therapy > Grade 1 if clinically relevant.
* Receiving medications or substances known to be strong inhibitors or inducers of CYP3A4.
* Any known intolerance to agents structurally similar to crizotinib.
* Congenital long QT syndrome or persistent corrected QT interval by Fredericia formula (QTcF) ≥ 500 msec.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 5 years
  Via RECIST 1.1
Progression-free survival | 5 years
  Via RECIST 1.1
Average Time-to-treatment Failure | 5 years
  Time from randomization to treatment discontinuation for any reason
Edmonton Symptom Assessment Scale (ESAS) Score | 5 years
  Patient related symptom improvement evaluated by ESAS
EQ5D-5L Questionnaire Score | 5 years
  Patient preference/health related utility evaluated by EQ5D-5L Questionnaire
Overall survival | 2 years
  Number of days from the date of randomization to the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Leighl, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada